CLINICAL TRIAL: NCT01537276
Title: Improve Hysterosalpingographic Accuracy by Real-time Fluoroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YiYang Zhu (Other)
Responsible Party: Sponsor-Investigator, YiYang Zhu, Center for reproductive medicine, Taizhou Hospital
Organization: Taizhou Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: taizhou201101
Record Dates: First submitted 2012-02-12; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Infertility
Keywords: hysterosalpingography; Fluoroscopy; diagnostic accuracy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- real-time fluoroscopy (Experimental): evaluating the tubal patency and pathology under fluoroscopy real-timely
  Interventions: Procedure: diagnose under real-time fluoroscopy
- respective image (No Intervention): evaluating the tubal patency and pathology by Two supine and two oblique static images.

INTERVENTIONS:
Procedure: diagnose under real-time fluoroscopy — radiologists evaluating the tubal patency under fluoroscopy real-timely.Findings of fluoroscopy were blind to the investigators when the static radiographs were re-analyzed by the same team of radiologists.
  Other Names: dynamic fluoroscopy
  Arms: real-time fluoroscopy

SUMMARY:
As an essential step of the infertile work-up, hysterosalpingogram (HSG) has some advantages including the lack of need for anesthesia, a non-invasive procedure with less cost and relative easy to put into practice. However, it would be failed to detect the extra-tubal and peritoneal pathology and would be also difficult to distinguish the obstruction caused by the spasm of intramural segment. Obviously, imaging quality plays a key role in diagnostic accuracy of the HSG, studies had taken four roentgenograms and combined with the fluoroscopy were reported a higher sensitivity and specificity than those only taken two images in the examination. And hybridized radiography with CT or MRI system may provide the good-quality of the HSG. It is also reported that the sonosalpingography (SSG), which detect the tubal patency in real time, can show pelvic pathologies better than HSG. However, no parallel study was designed to verify the hypothesis that combined the fluoroscopy and taken more images can improving the diagnostic quality of the HSG. The aim of this study is to evaluate whether the accuracy of HSG can be improved by real-time evaluating under the fluoroscopy.

DETAILED DESCRIPTION:
Tubal disease is responsible for 30-40% of female infertility in China. The lesions of fallopian tube include occlusion, hydrosalpinx, and adhesion. Many techniques were developed to assess the tubal pathology. Although laparoscopy can visualize the morphological abnormalities of fallopian tubes directly and is widely accepted as a gold standard for investigation of tubal patency, it is an invasive procedure and may carry of some risk. Hysterosalpingography, which uses contrast media and radiographic techniques to visualize the uterine cavity and tubal lumen, remains the first line screening since it was described by Carey.

As an essential step of the infertile work-up, HSG has some advantages including the lack of need for anesthesia, a non-invasive procedure with less cost and relative easy to put into practice. Additional, HSG may have a potential therapeutic effect with the use of oil soluble contrast media for examination. However, it would be failed to detect the extra-tubal and peritoneal pathology and would be also difficult to distinguish the obstruction caused by the spasm of intramural segment. In an early meta-analysis, HSG was regard as the limited use of evaluating the peritubal adhesions because of its low sensitivity. But in a recently small sample's report, the authors argued that the diagnostic accuracy of HSG in peritubal adhesion can be improved by analyzing some special signs on the radiographs.

Obviously, imaging quality plays a key role in diagnostic accuracy of the HSG, studies had taken four roentgenograms and combined with the fluoroscopy were reported a higher sensitivity and specificity than those only taken two images in the examination. And hybridized radiography with CT or MRI system may provide the good-quality of the HSG. It is also reported that the sonosalpingography (SSG), which detect the tubal patency in real time, can show pelvic pathologies better than HSG. However, no parallel study was designed to verify the hypothesis that combined the fluoroscopy and taken more images can improving the diagnostic quality of the HSG. The aim of this study is to evaluate whether the accuracy of HSG can be improved by real-time evaluating under the fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* women seeking for a infertility laparoscopy

Exclusion Criteria:

* acute low reproductive duct infection
* a known hypersensitivity to iodine
* genital bleeding or malignancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 263 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
diagnostic sensitivity, specificity, positive predictive value, negative predictive value of HSG in detecting tubal pathologies | participants will be followed by laparoscopy in 6 month after HSG
  The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) of HSG for diagnosis of tubal pathlogies. The pathlogies of tube is classified as the normal HSG, the proximal tubal obstruction, the hydrosalpinx (distal tubal obstruction), and the peritubal adhesions (at least one tube is patent) ,which is confirmed by laparoscopy in six month after HSG.

SECONDARY OUTCOMES:
diagnostic sensitivity, specificity, positive predictive value, negative predictive value of HSG in detecting tubal patency | participants will be followed by laparoscopy in 6 month after HSG
  The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) of HSG for diagnosis of tubal patency. The patency of tube is classified as two-sided occlusion, one-sided occlusion and two side patency,which is confirmed by laparoscopy in six month after HSG.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Zi Mao, MD, Study Director — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University
Locations (1):
- Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang, China